CLINICAL TRIAL: NCT05965895
Title: Ultrasound-Guided Continuous Serratus Anterior Plane Block Versus Intravenous Dexmedetomidine Infusion for Pain Control in Patients With Multiple Rib Fractures: A Prospective Randomized Clinical Trial.
Brief Title: Ultrasound-Guided Continuous Serratus Anterior Plane Block vs Dexmedetomidine Infusion in Patients With Rib Fractures.
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Dina Mahmoud Fakhry, Assistant Lecturer of Anesthesiology, Surgical Intensive Care and Pain Management, Beni-Suef University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FMBSUREC/09072023/Fakhry
Record Dates: First submitted 2023-07-20; First posted 2023-07-28 (Actual); Last update posted 2023-10-11 (Actual); Status verified 2023-10

CONDITIONS: Pain
Keywords: Serratus anterior; Dexmedetomidine; Rib; Fractures
MeSH Terms: conditions — Pain; Fractures, Bone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- US-guided SAP block group (Active Comparator): Patients will receive US-guided SAP block with a bolus of 2 mg/kg levobupivacaine made up to a volume of 40 ml followed by an infusion of 0.125% levobupivacaine will be commenced at rate of 8 ml/hr for 48 hr.
  Interventions: Procedure: Ultrasound-guided continuous serratus anterior plane block
- Dexmedetomidine group (Active Comparator): Patients will receive initial loading dose of dexmedetomidine of 1 µg/kg over 30 min followed by a continuous infusion at a rate of 0.5 µg/kg/hr for 48 hr.
  Interventions: Drug: intravenous dexmedetomidine infusion

INTERVENTIONS:
Procedure: Ultrasound-guided continuous serratus anterior plane block — Patients will receive US-guided SAP block with a bolus of 2 mg/kg levobupivacaine made up to a volume of 40 ml followed by an infusion of 0.125% levobupivacaine will be commenced at rate of 8 ml/hr for 48 hr.
  Other Names: Group S
  Arms: US-guided SAP block group
Drug: intravenous dexmedetomidine infusion — Patients will receive initial loading dose of dexmedetomidine of 1 µg/kg over 30 min followed by a continuous infusion at a rate of 0.5 µg/kg/hr for 48 hr.
  Other Names: Group D
  Arms: Dexmedetomidine group

SUMMARY:
The aim of this work is to compare analgesic efficacy in patients with multiple rib fractures who will be managed with Ultrasound-guided continuous serratus anterior plane block versus patients who will be managed with dexmedetomidine infusion.

DETAILED DESCRIPTION:
In thoracic trauma patients with rib fractures, the ability to cough and clear secretions is impaired by pain, leading to an increased risk of atelectasis, retention of secretions, chest infections and prolonged ICU stay thereby leads to significant morbidity, mortality and cost of treatment.Hence, aggressive pain management is a vital component of rib fracture management for the healing of rib fractures, improvement of pulmonary functions, and pulmonary rehabilitation.

The number of rib fractures >3, rib fracture locations, bilateral rib fractures, intraparenchymal pulmonary injuries, flail chest, and a first rib fracture influence the mortality rates.

The involvement of acute pain services in Multiple rib fractures (MRFs) is based on "Rib Fracture score". Rib fracture score = (breaks × sides) + age factor. "Breaks" is the total number of fractures to the rib. Score of 1 is for unilateral fractures and 2 for bilateral fractures. Age is factored into the equation due to an increased risk of complications (age factor = 0 if <50 years; 1 if 51-60 years; 2 if 61-70 years; 3 if 71-80 years; 4 if above 80 years). A score >7, requires the involvement of acute pain team.

There is a wide variety of strategies for treating acute pain , including multimodal opioid and non-opioid systemic analgesics, regional anesthesia including thoracic epidural analgesia (TEA), paravertebral blocks (PVB),intercostal nerve blocks and a recent expansion in the use of novel fascial plane blocks.

Ultrasound-guided Serratus Anterior Plane (SAP) block is an ultrasound (US) guided interfascial plane block which has been used in managing pain due to MRFs. It is a relatively recent technique, first described in 2013, that provides almost complete analgesia for the thoracic wall by blocking the lateral branches of the intercostal nerves from T2 to L2. Two planes were described, one superficial to serratus anterior muscle and second underneath the muscle and above the rib. It is a safe, simple to perform block with no significant contraindications or side effects. It can be performed in patients lying supine, rendering it particularly useful in polytrauma patients who are unable to sit up or turn lateral for regional blocks on the back. It can be safely given to polytrauma patients who may be having hemodynamic instability or coagulopathy, unlike epidural and paravertebral. There is a theoretical possibility of local anesthetic toxicity and hematoma such as other interfacial plane blocks. Pneumothorax is a potential complication, but under ultrasound guidance, it would be a remote possibility as the injection is far from the pleura between two muscles or above the rib.

Use of continuous techniques using catheters has the benefit of providing prolonged analgesia titrated to patient response.

Dexmedetomidine is a highly selective α-2 adrenoceptor agonist. It has sympatholytic, sedative, amnestic, and analgesic properties. It provides a unique analgesia, without respiratory depression best described as opioid- sparing. The analgesic properties of α-2 agonists are mediated by Supraspinal (locus ceruleus) and spinal (dorsal horn) mechanisms. Also it decreases sympathetic outflow through a central action in a dose-dependent manner, and these presynaptic sites of action are clinically significant because they modulate the release of norepinephrine. This inhibitory effect on neurotransmitter release is mediated by the blockage of calcium entry into nerve terminals. Systemic administration of the α-2 agonists has been tested in the perioperative period. The reduced opioid requirement was a feature of the administration of such group of medications. This feature is indirect evidence that these drugs have analgesic action. However, the perioperative period involves many conflicting factors. Clearly, the sedative effect may be the reason behind the reduced opioid requirements.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Rib fracture score of more than 7
* Patient with isolated multiple rib fractures, ●American Society of Anesthesiologists classification of physical status < IV
* Body mass index (BMI) ≤ 35.

Exclusion Criteria:

* Refusal of the patient
* Trauma survey include multiple injuries including head injuries, visceral and long bone fractures
* Intubated patients
* Known hypersensitivity to any study medication, ●Chronic opioid use or chronic pain patient, ●Hemodynamic instability
* Haemothorax or pneumothorax.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-08-01 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
Quality of analgesia measured by visual analogue scale | The first 48 hours.
  rate pain severity scored from 0 to 10; while 0 stands for no pain at all and 10 is the worst intolerable pain.

SECONDARY OUTCOMES:
parameters of adequate ventilation and oxygenation | at 1, 2, 3, 4, 8, 16, 24, 36, 48 hours.
  PaO2/FiO2 ratio and PaCO2 will be recorded
Sedation score | Every 8 hours for 48 hours
  Ramsay score was used to evaluate sedation. Score 1 represents agitated and uncomfortable patient. Score 2 represents cooperative and orientated patient. Score 3 represents a patient who can follow simple directions. Score 4 represents an asleep patient with a strong response to stimulation. Score 5 represents an asleep patient with a slow response to stimulation. Score 6 represents an asleep patient with no response to stimulation.

CONTACTS AND LOCATIONS:
Overall Officials: Dina M Fakhry, MD, Principal Investigator — Beni-Suef University
Locations (1):
- Beni-Suef University hospital, Banī Suwayf, Beni Suweif Governorate, Egypt